CLINICAL TRIAL: NCT04355325
Title: Randomized Controlled Clinical Trial to Compare Posterior Implant-Supported Modified Monolithic Zirconia and Metal-Ceramic Single Crowns: 5 Years Study
Brief Title: Posterior Implant-Supported Modified Monolithic Zirconia and Metal-Ceramic Single Crowns: 5 Years Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jordan University of Science and Technology (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Principal Investigator, Rola Abdelraheem Alhabashneh, Prof Rola Alhabashneh, Jordan University of Science and Technology
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Jordan
Record Dates: First submitted 2020-02-07; First posted 2020-04-21 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Posterior Occlusion; Fracture
Keywords: Implant; Zirconia; crown; molar
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: This single-blind split mouth study will enroll 60 participants, having to receive 120 dental Implants. They will be recruited from 3 dental centers in Jordan .
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Active Comparator): modified monolithic zirconia crowns At the time of the second optical impression, implants will be randomly allocated to either the test group (modified monolithic zirconia crowns) or the control group (metal ceramic crowns), using a computer-generated randomization list.
  Interventions: Device: modified monolithic zirconia crowns; Device: Metal Ceramic crowns
- control (Placebo Comparator): metal ceramic crowns At the time of the second optical impression, implants will be randomly allocated to either the test group (modified monolithic zirconia crowns) or the control group (metal ceramic crowns), using a computer-generated randomization list.
  Interventions: Device: modified monolithic zirconia crowns; Device: Metal Ceramic crowns

INTERVENTIONS:
Device: modified monolithic zirconia crowns — outcomes and complications of implant restoration
  Other Names: Zirconia
Device: Metal Ceramic crowns — outcomes and complications of implant restoration
  Other Names: Metal-Ceramic

SUMMARY:
The outcome of implant therapy has been presented in the majority of clinical studies by focusing only on implant survival without providing detailed information on the reconstructions . However, for decision making, it is important to know the survival rates and the incidence of biological and technical complications not only for the implants but also for the reconstructions. Thus, the selection of restoration materials should be based on proper optical characteristics in addition to biocompatibility and sufficient strength of materials.

Monolithic zirconia has been used in posterior region, especially for single crowns, in order to eliminate the veneer cracking, But Since monolithic zirconia are relatively new, few randomized, controlled clinical studies have evaluated their success. There is only one study identified regarding the performance of monolithic ceramic restorations bonded to Ti inserts, investigating the clinical outcome of using monolithic or modified monolithic zirconia implant-supported single crowns and comparing outcomes and complications of metal-ceramic and monolithic or modified monolithic zirconia implant supported single crowns.

More clinical studies to evaluate the performance of CAD/CAM monolithic implant-supported restorations bonded to Ti inserts and bases and compare their survival, success and complication rates with other restorative options [with a mean follow-up period of at least 5 years are required for a meaningful interpretation of the survival and complication rate .

So this study aims to investigate outcomes and complications of implant supported modified monolithic zirconia and metal-ceramic single crowns in the posterior region of the mouth.

The null hypothesis is that there is no difference between modified monolithic zirconia and metal-ceramic posterior implant-supported SCs in prosthetic complication rates.

DETAILED DESCRIPTION:
Background: Dental implants restored with single crowns (SCs) have been reported to have a comparable survival rate and fewer technical complications compared to multiple-unit implant-supported FDPs. Porcelain-fused to metal restorations were the golden standard option for implant supported reconstructions in the past, but nowadays, the application of all-ceramic restorations in general and specifically zirconia as a restorative material for implant-supported single crowns has increased utilizing the CAD/CAM technology. The continuous technological progress in both the computer-based development and the dental manufacturing process ensures new opportunities in the clinical workflow. A fully digital pathway in a model-free approach or a combination of these workflows is now possible.

Purpose: The purpose of this randomized controlled clinical trial is to investigate the prosthetic outcomes of posterior implant-supported single crowns (SCs) with a modified monolithic zirconia or metal-ceramic design utilizing the digital workflow at 1, 3 and 5 years of loading.

Materials and methods: This single-blind split mouth study will enroll 60 participants, having to receive 120 dental Implants. They will be scheduled for a bilateral posterior single-unit prosthetic rehabilitation supported by one implant in the posterior region of the maxilla or the mandible (premolars, molars). A fully digital pathway will be followed. A CT scan will be performed without any template. An intraoral optical impression using CEREC Omnicam scanner will be made. A virtual set-up of the prosthetic reconstruction, as well as a surgical template with optimal 3-D implant positioning will be designed then printed using a 3-D printer without the need of any physical model. Straumann bone level implants with either a wide diameter (Ø4.8 mm) or regular diameter (Ø4.1 mm) with a minimum length of 8 mm will be inserted. Implants will be loaded after 3 months of submerged healing. A second intraoral optical impression will be made using CEREC Omnicam scanner and Straumann scanbody. The implant-supported prosthetic suprastructure will be designed. Implants will be randomly allocated to either the test group modified monolithic zirconia crowns (MMZ) or the control group metal ceramic crowns (MC), using a computer-generated randomization list. A digital model with movable dies will be 3-D printed, then used to adjust restoration in terms of occlusal and proximal contacts. Prefabricated screw-retained Titanium abutments (Variobase Abutment; Straumann) will be used as the metal substructures of the crowns and will be secured to lab analogues on the digitally printed casts. Metal/ zirconia substructures with a hole for the screw retention will be designed using the CAD software and will be anatomically reduced by 1 mm to allow for porcelain veneering then will be laser-printed/ dry milled. Hand layering of glass ceramic will be made on the surface. Crowns will be cemented extraorally to titanium abutments using dual cure resin cement to make one-piece screw-retained single crown. The screw-retained single crowns and titanium abutments will be inserted intraorally with 35 Ncm torque and screw-access holes will be restored with Teflon and light-polymerized composite resin. The implant-supported SCs will be examined after 1, 3 and 5 years for survival and technical complications.

Clinical significance: to evaluate the survival and prosthetic complication rates of zirconia-ceramic and metal-ceramic implant-supported single crowns at 1, 3 and 5 years of service. In addition to that, the digital workflow for implant supported single crowns will be evaluated for efficiency, accuracy, time and cost compared to conventional workflow.

ELIGIBILITY:
Inclusion Criteria:

* · Participants will be required to sign informed consents prior to inclusion in the study.

  * Aged between 21 to 55 years, with no contraindications to dental treatment.
  * Need implant supported single crown in the maxillary and/or mandibular premolar and/or molar area
  * No systemic disease.
  * No signs of bruxism.
  * Full-mouth plaque scores and full-mouth bleeding scores of <25%
  * Good overall dental health, no active caries, no active periodontal disease, and periodontal pocket depths not greater than 4 mm.
  * Adequate bone height and width at areas of proposed implant sites
  * Adequate interocclusal distance to accommodate the prosthesis
  * Space width with mesial -distal width of at least 6 mm.
  * Good oral hygiene and compliance with oral hygiene instructions as determined by the amount of plaque present on tooth surfaces
  * Thick or medium gingival biotype.
  * Bilateral one missing tooth being a premolar or molar in the maxilla or mandible with adjacent natural teeth.
  * Fixed teeth opposing the edentulous area and a full complement of teeth or restored teeth in all other areas.

Exclusion Criteria:

* Systemic disease

  * Pregnant and lactating women
  * Unwilling to receive radiographs
  * Presence of clinically active periodontal disease as expressed by probing pocket depths 4 mm in combination with bleeding on probing
  * Presence of peri-apical lesions or any other abnormalities in the region as detected on a radiograph.
  * Subjects that get diagnosed with any systemic disease, start smoking, or become pregnant during the study period will be excluded from the study

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-02 (Actual); Primary Completion 2024-05-02 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
Screw loosing | 5 years
  Alpha rating: no screw loosening Bravo rating: loose screw that can be retightened Delta rating: fractured screw that needs replacement
Marginal integrity | 5 years
  Visual inspection with dental explorer to the abutment-restoration interphase under fourfold to fivefold optical magnification. Digital bitewing radiographs with standardized paralleling technique using Ring holders and analogue films will be taken at baseline then at each recall visit and compared together for any misfits or gaps. Alpha rating: no visible or soundable gap Bravo rating: marginal gap slightly soundable Charlie rating: explorer penetrates a significant crevice Delta rating: restoration needs to be replaced
chipping of veneering ceramic | 5 years
  Visual and tactile inspection of the restorations will be made to check for any chippings of the restoration. Fourfold to fivefold optical magnification will be used. Clinical photographs will be taken for crowns and neighboring teeth at delivery stage. Impressions will be made as well and poured into stone. New impressions will be made at each recall visit, poured into stone, then stone casts will be evaluated using a light microscope and compared with surface topography of casts made at prosthetic delivery stage to detect any potential minor chip-off fractures.
  * Alpha rating: No fracture
  * Bravo rating: minor chipping (polishable)
  * Charlie rating: major chipping (up to framework)
  * Delta rating: restoration needs to be replaced If chipping rating changes during the observation period, the most severe rating will be recorded
occlusal roughness | 5 years
  Crowns will be dried at each recall visit and visually inspected under fourfold to fivefold optical magnification for any roughness. Alpha rating: no roughness Bravo rating: slight roughness (< 2mm) Charlie rating: obvious roughness (> 2mm) Delta rating: restoration needs to be replaced If roughness rating changes during the observation period, the most severe rating will be recorded
framework fracture | 5 years
  Visual and tactile inspection of the restorations will be made to check for fracture or loss of the restoration. Fourfold to fivefold optical magnification will be used. Clinical photographs will be also taken for crowns and neighboring teeth at delivery stage then at each recall visit and compared together.
  * Alpha rating: No fracture
  * Delta rating: restoration needs to be replaced If fracture rating changes during the observation period, the most severe rating will be recorded.

SECONDARY OUTCOMES:
Marginal bone loss: | 1 year
  Digital bitewing radiographs with standardized paralleling technique using Ring holders and analogue films will be taken at the days of implant placement, at baseline, at 6, at 12 months, then at each recall visit and compared together for marginal bone loss
Crown de-bonding | 5 years
  Tactile inspection for any loosening of the restoration. History taking from the patient for any incidence of crown loosening, movement upon eating or complete separation from underlying abutment. Alpha rating: no crown de-bonding Bravo rating: crown de-bonding that can be re-bonded Delta rating: de-bonded crown that needs replacement

CONTACTS AND LOCATIONS:
Overall Officials: Rola Alhabshneh, Prof, Principal Investigator — JUST
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No